CLINICAL TRIAL: NCT00245752
Title: Randomised Study of the Effect of Acupuncture as Induction of Labour
Brief Title: Can Acupuncture be Used as Preparation for Induction of Labour
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Skejby Research Fond (Unknown); Ringkjøbing County Research Fond (Unknown); Union of Midwives Research Fond (Other)
Responsible Party: Jette Modlock, Skejby Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20040001
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Pregnancy Overdue - Week 41+6
Keywords: post term pregnancy; acupuncture; induction
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): in points bilaterally inBL 67, LI 4, SP6, one in GV20.
  Interventions: Device: acupuncture
- 2 (Sham Comparator): sham acupuncture
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — acupuncture in points bilaterally: BL 67, LI 4, SP6, one in GV20.
  Other Names: Seirin Steel needles; and Park Sham needles

SUMMARY:
The purpose of the study is to evaluate whether acupuncture can be used to ripen cervix before medicinal induction of labor or even be used as method for induction, and thereby eliminating other and more potentially harmful methods.

DETAILED DESCRIPTION:
Acupuncture has become a natural part of the range of treatments in obstetric departments in Denmark, but there is only little evidence to the effect of acupuncture.

Many of the induction procedures currently in use in Denmark also have a little risk of side effects. to mention a few: There is a increased risk of maternal and neonatal infection, bleeding, ruptured membranes and placental disruption as result of the use of endocervical balloon catheter. In connection with manual rupture of membranes there is an increased risk of umbilical prolapse, maternal and neonatal infection, affected fetal heart rate, scratches on the scalp and placental bleeding. By using misoprostol there has been seen hyperstimulation of uterus causing affected fetal heart rate.

Many women are asking for alternatives to the existing methods used in obstetric dept.s.

In order to assess the effect, or lack of, acupuncture might have, we want to use acupuncture in the study group on acupuncture points on hands, feet, ankles and back of the head. The control group will get placebo acupuncture needles on same locations. The included women will be treated with the kind of acupuncture that counts for the group to which shes been allocated on gestational age 41+6 at 8:00 am and 2:30 pm.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 41+6
* Normal pregnancy, expecting a healthy baby
* Verified due date

Exclusion Criteria:

* Women who do not speak or understand Danish
* Multiple pregnancy
* In active labour
* Previous sectio
* Maternal diseases (i.e. Diabetes, preeclampsia, heart diseases)
* Fetal diseases (i.e. foetus mors, IUGR, hydrocephalus)
* Previous complicated delivery i.e. low Apgar score
* Allergic to metal
* Anticoagulatory treatment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
In active delivery or not (over or equal to 3 cm) | 24 hrs

SECONDARY OUTCOMES:
Degree of dilatation of orificium | 24 hrs
Ruptured membranes or not, | 24 hrs
Increase in uterine activity or not, | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Niels Uldbjerg, Professor, Principal Investigator

REFERENCES:
- [Derived] Modlock J, Nielsen BB, Uldbjerg N. Acupuncture for the induction of labour: a double-blind randomised controlled study. BJOG. 2010 Sep;117(10):1255-61. doi: 10.1111/j.1471-0528.2010.02647.x. Epub 2010 Jun 24. PMID 20573151